CLINICAL TRIAL: NCT02583646
Title: Investigating the Impact of Obesity on Pubertal Development in Girls
Status: Recruiting | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160006; 16-E-0006
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-08

CONDITIONS: Obesity; Puberty; Normal Physiology
Keywords: Obesity; Puberty; Ultrasound; Pediatric; Natural History
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal weight: Girls age 8-14 below 85% in respect to weight for their age group
- overweight: Girls age 8-14 at or above 85% in respect to weight for their age group

SUMMARY:
Background:

Studies suggest that overweight girls may be developing breast tissue, and therefore starting puberty, earlier than normal weight girls. However, it is hard to distinguish breast tissue from fatty tissue. Researchers think that by using breast ultrasound, among other tests, they can do a better job of telling whether an overweight girl has breast tissue. This will help them understand if overweight girls are truly entering puberty before normal weight girls.

Objective:

To find out if overweight girls go through puberty earlier than normal weight girls.

Eligibility:

Healthy girls 8-14 years old who:

* Are normal weight or overweight
* Have some breast development
* Have not started their first period

Design:

Parents of participants will be screened over the phone.

Most participants will have 1 visit. However, they can choose to have multiple visits within 4 weeks. The visit will include:

* Physical exam that includes examination of the breasts and genital area
* Breast ultrasound: A small hand-held device will be passed back and forth over the chest. It uses sound waves to create a picture of the breast tissue.
* Pelvic ultrasound: A small, handheld device will be passed back and forth over the lower belly. It uses sound waves to create a picture of the ovaries.
* Urine and blood test
* A special x-ray called a DXA to measure the amount of fat in the body: The participant will lie still on a table while the x-ray takes pictures of the body.

X-ray of the hand: The picture will tell researchers how mature the participant s bones are.

Participants may be asked to come back 6 months later to repeat these tests.

...

DETAILED DESCRIPTION:
Over the past decade, there has been an alarming trend toward earlier breast development in girls. The contemporaneous obesity epidemic has led to speculation that obesity may be driving early puberty. However, questions remain about the validity of reports of early puberty among obese girls due to the difficulty in distinguishing fatty tissue from breast tissue in this population. The physiological basis for early puberty among obese girls is also unknown. The current proposal aims to investigate pubertal development in pre-menarchal obese compared with normal weight girls using more robust methods such as breast morphological staging via ultrasonography and intensive reproductive axis phenotyping. Study procedures include blood draws, DXA (for body composition), hand x-ray (for bone age), breast and transabdominal (pelvic) ultrasounds, and anthropometrics.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Girls without a chronic medical condition
* Normal weight (BMI 5th-85th%) or overweight/obese (BMI > 85th%)
* 8-14 years old
* Some breast development
* Pre-menarchal

EXCLUSION CRITERIA:

* Treated with medications that may affect reproductive hormones (e.g. birth control pills).
* Pregnancy

During the study, the PI s discretion may be used to determine final eligibility. The PI s discretion may be used at any point in the study (pre-screening, clinical/lab assessments, etc.) to ensure participants are not subjected to unnecessary procedures or visits.

Ages: 8 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-12-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
To determine the correlation between Tanner breast staging and breast maturation scores using breast ultrasound in girls | semiannually
  To test the hypothesis that breast maturation in obese and normal weight girls primarily reflects hypothalamic-pituitary-ovarian activation as opposed to local (breast adipose tissue) estrogen production, we will use linear regression to determine if the relationship between breast maturation and ovarian size, uterine size and bone age (all markers of end organ response to estrogen) differs between the two weight groups (group by ovarian/uterine size/bone age interaction term). The finding of similar regression lines in the two groups would support this hypothesis while an upward shift in the regression line (greater y-intercept, similar slope) in the obese girls would indicate that a given breast maturation stage is achieved at a smaller ovarian/uterine volume and younger bone age in obese girls, suggesting the presence of an additional source of estrogen (adipose tissue) in obese girls.

SECONDARY OUTCOMES:
To determine the contribution of peripheral aromatization to breast development in obese girls. | semiannually
  Repeated measures from the same subject (visits 1,2, and follow up visits) will provide preliminary data for future studies investigating whether there is a difference in the pace of pubertal development in obese compared with normal weight girls. Squamous cells in the urine sample will be categorized as either superficial (mature; eg indicating estrogen exposure) or other . The primary measure of estrogenization will be the percent of superficial cells (%S), as previously described (Adgent 13, Robine 88). The %S will be compared between normal weight and obese subjects after controlling for breast stage determined by ultrasound. We anticipate that up to 25% of urine specimens may need to be excluded because of insufficient cells or inflammation and this may require an increase in enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie D Shaw, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS, Research Triangle Park, Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herman-Giddens ME, Kaplowitz PB, Wasserman R. Navigating the recent articles on girls' puberty in Pediatrics: what do we know and where do we go from here? Pediatrics. 2004 Apr;113(4):911-7. doi: 10.1542/peds.113.4.911. No abstract available. PMID 15060243
- [Background] Kaplowitz PB. Link between body fat and the timing of puberty. Pediatrics. 2008 Feb;121 Suppl 3:S208-17. doi: 10.1542/peds.2007-1813F. PMID 18245513
- [Background] Ahmed ML, Ong KK, Dunger DB. Childhood obesity and the timing of puberty. Trends Endocrinol Metab. 2009 Jul;20(5):237-42. doi: 10.1016/j.tem.2009.02.004. Epub 2009 Jun 21. PMID 19541497
- [Derived] Ortega MT, McGrath JA, Carlson L, Flores Poccia V, Larson G, Douglas C, Sun BZ, Zhao S, Beery B, Vesper HW, Duke L, Botelho JC, Filie AC, Shaw ND. Longitudinal Investigation of Pubertal Milestones and Hormones as a Function of Body Fat in Girls. J Clin Endocrinol Metab. 2021 May 13;106(6):1668-1683. doi: 10.1210/clinem/dgab092. PMID 33630047
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-E-0006.html